CLINICAL TRIAL: NCT03277092
Title: Impact of Near Infrared Light in Paediatric Blood Drawing Centre on Rate of First Attempt Success and Time of Procedure
Brief Title: Near Infrared Light in Paediatric Blood Drawing Centre
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC 22/17
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-06

CONDITIONS: Blood Drawing Procedure
Keywords: Child, blood drawing procedure, near Infrared light

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VeinViewer® group (Experimental): Use of near infrared light to perform blood draw (VeinViewer®)
  Interventions: Device: VeinViewer®
- Usual care group (Active Comparator): Blood drawing performed traditionally
  Interventions: Procedure: Usual care

INTERVENTIONS:
Device: VeinViewer® — Near-infrared (NIR) technology consists on light-emitting diodes placed underneath the hand, that makes vessels visible by projecting the processed image in a green light directly on to the puncture site
  Arms: VeinViewer® group
Procedure: Usual care — The blood drawing is performed traditionally
  Arms: Usual care group

SUMMARY:
Reaching a peripheral venous access or making a blood sample in a scared infant or toddler can be challenging even for experienced nurses o pediatricians. Up to 60% of children report pain and distress during venipuncture and multiple attempts can result in more difficult physical and emotional conditions for subsequent insertions so that the procedure should be performed with the less number of punctures as possible. In about one third of children, more than one attempt is required to achieve peripheral intravenous cannulation. In the last years, specific tools have been developed to enhance the success in venipuncture or incannulation. Near-infrared (NIR) technology consists on light-emitting diodes placed underneath the hand, that makes vessels visible by projecting the processed image in a green light directly on to the puncture site. According to previous studies, NIR had shown a trend in reduction of time employed for a blood sample, in children younger of 6 yr.

The aim of this trial is to investigate if the use of the VeinViewer® in a pediatric blood drawing center could decrease time spent to perform the procedure and improve the rate of first attempt success.

ELIGIBILITY:
Inclusion Criteria:

* subjects accessing the outpatient blood-drawing service

Exclusion Criteria:

* application of topical anaesthetic cream

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 115 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Time to perform the procedure | Intraprocedural
  In seconds, from the placement of the tourniquet until the blood flows in the needle

SECONDARY OUTCOMES:
Success at first attempt | Intraprocedural
  Percentage of success at first attempt

CONTACTS AND LOCATIONS:
Overall Officials: Egidio Barbi, MD PhD, Principal Investigator — IRCCS Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Conversano E, Cozzi G, Pavan M, Minute M, Gortan E, Montico M, Vecchi Brumatti L, Ronfani L, Barbi E. Impact of near infrared light in pediatric blood drawing Centre on rate of first attempt success and time of procedure. Ital J Pediatr. 2018 May 25;44(1):60. doi: 10.1186/s13052-018-0501-1. PMID 29801519